CLINICAL TRIAL: NCT05824429
Title: Effects of Connective Tissue Manipulation on Clinical Symptoms and Pelvic Floor Muscle Functions in Children With Lower Urinary Tract Dysfunction
Brief Title: Connective Tissue Manipulation on Pelvic Floor Muscle Functions in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Collaborators: Tugtepe Pediatric Urology Clinic (Other)
Responsible Party: Principal Investigator, Melis ünal, Physiotherapist, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MelisU
Record Dates: First submitted 2023-04-05; First posted 2023-04-21 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Pelvic Floor; Urinary Incontinence; Connective Tissue
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connective Tissue Manipulation Group (Experimental): Urotheraphy Diaphragmatic Breathing Exercises Pelvic Floor Muscle Exercise Connective Tissue Manipülation
  Interventions: Other: Urotherapy; Other: Diaphragmatic Breathing Exercises; Other: PFM Exercises; Other: Connective Tissue Manipulation
- Control Group (Active Comparator): Urotheraphy Diaphragmatic Breathing Exercises Pelvic Floor Muscle Exercise
  Interventions: Other: Urotherapy; Other: Diaphragmatic Breathing Exercises; Other: PFM Exercises

INTERVENTIONS:
Other: Urotherapy — Urotherapy is an umbrella term that includes components such as information about bladder function and problem, lifestyle changes including the regulation of voiding and fluid intake times, correct toilet positions, information about bladder irritants, and motivation. All participants included in our study will be given urotherapy training before starting PFM exercises and CTM with their families.
Other: Diaphragmatic Breathing Exercises — In our research, diaphragm breathing exercises will be applied to both groups before starting PFM exercises in sessions for 8 weeks, 3 days a week.
Other: PFM Exercises — PFM exercises will be started after children learn to contract and relax their PFM in isolation without the use of auxiliary muscles. In the exercises, fast and slow contractions targeting type 1 and type 2 muscle fibers will be taught to increase both strength and endurance of PFM.
Other: Connective Tissue Manipulation — CTM is a reflex treatment technique that is applied manually by physiotherapists to the skin area and acts on some cells and connective tissue by making short and long pulls (. In our study, CTM will be applied to our study group, where CTM and PFMR will be applied together, 3 days a week, for a total of 8 weeks.
  The application will be made to the basic region (sacral), lower thoracic, abdominal and anterior pelvic region.
  Arms: Connective Tissue Manipulation Group

SUMMARY:
Lower urinary tract dysfunction (LUTD) is a disease group with subgroups that make up 40% of the patients were admitted to the pediatric urology clinic. The treatment of LUTD includes pharmacological, surgical treatment, neuromodulation, urotherapy, and pelvic floor muscle training. Conservative methods include bladder training, changing lifestyle and eating habits, pharmacological treatment, and physiotherapy approaches.

Physiotherapy approaches used in the treatment of LUTD are; biofeedback, electrical stimulation applications, diaphragm breathing exercises, and manual therapy methods.

The aim of our study is to compare the effects of Connective Tissue Manipülation (CTM) , which will be applied in addition to Pelvic Floor Muscle Rehabilitation (PFMR) for 8 weeks, on LUTD symptoms, pelvic floor muscle functions, uroflowmetry values and quality of life compared to PTMR applied alone for 8 weeks in children with LUTD.

DETAILED DESCRIPTION:
LUTD is clinical without any neuropathy; It refers to conditions that occur with symptoms such as urinary incontinence, urgency, increased or decreased urination during the day, dysuria, difficulty in starting to void, and the feeling of not being able to empty the bladder adequately.

Pelvic floor muscles (PFM) are known to be involved in the pathophysiology of LUTD. PFM needs to function normally during both the storage and voiding phase. In the literature, there are studies with positive results using PFM exercises in the treatment of symptoms in children with LUTD.

Connective Tissue Manipulation (CTM) can also be used within the scope of physiotherapy approaches that can be applied in children with LUTD. CTM is a reflex treatment technique that is applied manually by physiotherapists to the skin area and acts on some cells and connective tissue by making short and long pulls. Although the mechanism of action of CTM has not been fully elucidated, it is known to reduce organ dysfunctions by maintaining the balance between the parasympathetic and sympathetic components of the autonomic nervous system through segmental and supra-segmental cutaneous reflex pathways.

We think that CTM applied in addition to PFMR in the pediatric population can reduce LUTD symptoms by restoring the autonomic nervous system balance and increasing vascularity in the bladder. Therefore, the aim of our study is to compare the effects of CTM, which will be applied in addition to PFMR in children with LUTD, on LUTD symptoms, pelvic floor muscle functions, uroflowmetry values, and quality of life compared to PTCR applied alone.

ELIGIBILITY:
Inclusion Criteria:

* Be in the age range of 5-15 years
* Diagnosed with LUTD by a pediatric urologist according to the criteria set by the ICCS
* Volunteering by parent and child to participate in the study

Exclusion Criteria:

* Having any problems of neurogenic origin
* Any condition that affects the ability of the parent or child to respond to the scales to be used (mental retardation, cognitive problems, etc.)
* Malformations or anatomical differences in the urinary system
* Participants who discontinued treatment
* Presence of a urological surgery history
* Being on medication
* Having constipation and/or fecal incontinence

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2023-07-05 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
EMG- Uroflowmetry | 8 weeks
  In the uroflowmetry evaluation to be applied in our study, in case the patient's urge to urinate occurs, urination will be requested into the AYMED® brand EMG uroflowmetry container with a sensor system.
Pelvic Floor Muscle Activation Assestment | 8 weeks
  In our study, the PTM activation values of the participants will be measured by the physiotherapist before and after the treatment using the NeuroTrac Myoplus4 Pro device.
Bladder Diary | 8 weeks
  Thanks to the diary, parameters such as the child's daytime voiding frequency and volume, the amount and type of fluid taken, the duration of voiding, the presence of a sense of urgency, and the degree of urinary incontinence can be evaluated.In our study, the parents of the children will be trained by the physiotherapist to fill the bladder diary correctly, and they will be asked to fill in the 48-day voiding chart
Dysfunctional Voiding and Incontinence Scoring System (DVISS) | 8 weeks
  It is a questionnaire that evaluates the severity of lower urinary tract dysfunctions and is completed by parents. DVISS questions for all participants before and after the treatment will be filled by the physiotherapist by reading each question to the parents one by one.
Clinical Symtoms Information Form | 8 weeks
  Clinical symptoms will be recorded by the pediatric urologist by asking questions to the families and children and taking a detailed history during the face-to-face interview.

SECONDARY OUTCOMES:
Post-Voiding Residue (PVR) | 8 weeks
  With pelvic ultrasound, the bladder volume, the amount of urine in the bladder before voiding and the amount of urine remaining in the bladder after voiding can be evaluated.
Pediatric Incontinance Questionnaire (PinQ) | 8 weeks
  Bower et al. developed the PinQ scale in 2005 for use in children with urinary incontinence.In our study, the PinQ scale will be filled in by the physiotherapist before and after the treatment by reading each question to the children one by one.
Connective Tissue Evaluation | 8 weeks
  In our study, the responses of connective tissue inspection,palpation and circulation will be evaluated by examining both before and after treatment in the group in which PFMR will be applied only with CTM.

CONTACTS AND LOCATIONS:
Overall Officials: Halil Tuğtepe, Prof Dr, Study Chair — Tugtepe Pediatric Urology Center; Melis Ünal, PT, Study Director — Tugtepe Pediatric Urology Center
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No